CLINICAL TRIAL: NCT05733260
Title: A Resistance Training Program for Black Women: Project F.I.R.E.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Danielle D Wadsworth, Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-492 FB
Record Dates: First submitted 2022-12-16; First posted 2023-02-17 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally Tailored (Experimental): 10 weeks of resistance training utilizing culturally tailored prompts, feedback and high autonomy approaches.
  Interventions: Behavioral: Exercise
- Control (Experimental): 10 weeks of resistance training
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 10 weeks of resistance training.

SUMMARY:
This study will utilize a randomized control trial design, with participants randomly assigned to a theoretically-based culturally tailored intervention or standard of care group. Baseline (Week 0), 12-week, and 3-month follow-up (Week 24). Body composition and adherence will be tracked throughout the study. The exercise intervention will include a total body resistance training protocol and will take place at local fitness center. Participants will be randomized to either the theoretical-based culturally tailored intervention group or the standard exercise group in which each will be facilitated and supervised by a Black-trained research personnel following culturally tailored recommendations. All participants will attend a 10-week resistance training program twice per week for a total of 20 sessions from Weeks 2-11. Week 1 will be used to familiarize the participants with the resistance training exercises. Those randomized to the culturally tailored intervention group will receive health education, weekly text messages and self-regulatory strategies to overcome barriers to exercise. Participants will return for post testing at weeks 12 and 24.

DETAILED DESCRIPTION:
This study will utilize a randomized control trial design, with participants randomly assigned to a theoretically-based culturally tailored intervention or standard of care group. Baseline (Week 0), 12-week, and 3-month follow-up (Week 24). Body composition and adherence will be tracked throughout the study. The exercise intervention will include a total body resistance training protocol and will take place at local fitness center. Participants will be randomized to either the theoretical-based culturally tailored intervention group or the standard exercise group in which each will be facilitated and supervised by a Black-trained research personnel following culturally tailored recommendations. All participants will attend a 10-week resistance training program twice per week for a total of 20 sessions from Weeks 2-11. Week 1 will be used to familiarize the participants with the resistance training exercises. Those randomized to the culturally tailored intervention group will receive health education, weekly text messages and self-regulatory strategies to overcome barriers to exercise. Participants will return for post testing at weeks 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 34 years
* Identify as a black female
* Not actively participating in some type of exercise on a regular basis (at least three days a week for the past three months)
* Low risk for medical complications from exercise (as determined by the PAR-Q),
* Not pregnant or planning to become pregnant throughout the duration of the study
* Must live, work, or be a student in the city of Auburn, AL

Exclusion Criteria:

* women over 35
* Women who do not identify as black
* Regular exercisers,
* Pregnant women
* Women who do not have residency within Auburn AL

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Body Composition | 12 weeks
  Changes in body fat percentage assessed by dual x-ray absorptiometry
Body Composition | 24 weeks
  Changes in body fat percentage assessed by dual x-ray absorptiometry

SECONDARY OUTCOMES:
Adherence to resistance training | 12 weeks
  The number of days resistance training is completed each week.
Adherence to resistance training | 24 weeks
  The number of days resistance training is completed each week.

IPD SHARING:
Plan to Share IPD: No